CLINICAL TRIAL: NCT00004928
Title: A Phase I Study of 1,25 Dihydroxy-Vitamin D3 (Calcitriol) in Patients With Prostate Cancer
Brief Title: Calcitriol and Zoledronate in Treating Patients With Progressive Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-073; CDR0000067612 (Registry Identifier: PDQ (Physician Data Query)); NCI-H00-0048
Record Dates: First submitted 2000-03-07; First posted 2003-05-14 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; Zoledronic Acid

INTERVENTIONS:
Dietary Supplement: calcitriol
Drug: zoledronic acid

SUMMARY:
RATIONALE: Calcitriol may help prostate cancer cells develop into normal cells. Zoledronate may delay or prevent the formation of bone metastases. Combining calcitriol and zoledronate may be an effective treatment for progressive prostate cancer.

PURPOSE: Phase I trial to study the effectiveness of combining calcitriol with zoledronate in treating patients who have progressive prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of calcitriol administered with zoledronate in patients with progressive prostate cancer.
* Assess the effects of this regimen on calcium homeostasis and bone turnover in this patient population.
* Assess changes in PSA in patients treated with this regimen.
* Determine other antitumor effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study of calcitriol.

Patients receive oral calcitriol weekly for 3 consecutive days and zoledronate IV monthly. Treatment continues in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of calcitriol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prior localized adenocarcinoma of the prostate that has undergone definitive radiation or surgery and demonstrates progression biochemically with all of the following:

  * Baseline PSA at least 4 ng/mL
  * At least a 50% increase in PSA over at least 3 determinations taken at more than 2 week intervals
  * No radiographically evident disease
  * Neoadjuvant hormonal therapy prior to radical prostatectomy or radiotherapy allowed
  * Treatment in an intermittent approach allowed if off therapy for at least 12 weeks OR
* Histologically confirmed androgen-independent adenocarcinoma of the prostate with all of the following:

  * Progression on primary hormonal treatment (e.g., orchiectomy, estrogen therapy, gonadotropin-releasing hormone analog with or without an antiandrogen) with either new osseous lesions in bone, a greater than 25% increase in bidimensionally measurable tumor mass, or rising PSA values (rising PSA on any 3 determinations taken at at least weekly intervals, to greater than 50% above baseline PSA) despite castrate levels of testosterone (no greater than 30 ng/mL)
  * If receiving antiandrogen as part of primary hormonal therapy, must meet criteria above for progression after discontinuation of antiandrogen
  * No change in hormonal therapy (including prednisone or dexamethasone) within the past 2 weeks
  * If no prior surgical orchiectomy, must continue on medical therapies to maintain castrate levels of testosterone
  * Prior chemotherapy, palliative radiotherapy, or radioisotope treatment allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL OR
* SGOT less than 3 times upper limit of normal

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No history of nephrolithiasis
* Must have 2 functioning kidneys

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Pulmonary:

* No severe debilitating pulmonary disease

Metabolic:

* No pre-existing endocrine or metabolic disorders that impact calcium regulatory axis including hypercalcemia (ionized serum calcium greater than 5.3 mg/dL or total calcium greater than 10.5 mg/dL) or hypercalciuria (greater than 300 mg urinary calcium/24 hours)

Other:

* No active secondary malignancy except nonmelanoma skin cancer
* Must maintain low calcium diet (less than 800 mg calcium daily)
* No uncontrolled serious active infection
* No history of malabsorption disorders
* No history of inflammatory bowel disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* Recovered from prior endocrine therapy

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy to sole measurable lesion

Surgery:

* See Disease Characteristics
* Recovered from prior surgery
* No concurrent surgery to sole measurable lesion

Other:

* No other concurrent cholecalciferol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States